CLINICAL TRIAL: NCT05555004
Title: Evaluation of Probiotic (L.Reuteri) Survival in Presence of Prebiotic Galacto-oligosaccharides
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Based on slow recruitement and Interim analysis recommendation, the core team decide to stop the study
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2113NR
Record Dates: First submitted 2022-07-14; First posted 2022-09-26 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: comparator-controlled
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TEST1 (Experimental)
  Interventions: Other: TEST1
- TEST2 (Experimental)
  Interventions: Other: TEST 2

INTERVENTIONS:
Other: TEST1 — Toddler milk with preconditioned L. reuteri and containing GOS
  Arms: TEST1
Other: TEST 2 — Toddler milk with standard/non-preconditioned L. reuteri and not containing GOS.
  Arms: TEST2

SUMMARY:
This research study will compare the effect of test product #1 (containing a probiotic with the Galacto-OligoSaccharides fiber. GOS) and test product #2 (containing a probiotic without the GOS fiber) to understand how they can contribute to healthy digestion in toddlers between the age of 24 - 36 months. The hypothesis is that L. reuteri from TEST#1 will demonstrate an improved survival in the GIT of toddlers compared to that of TEST#2.

This study is a single-centre, randomized, double-blind, comparator-controlled, parallel group study. The study will be conducted at the Clinical Innovation Lab (CIL) at Nestlé Research.

ELIGIBILITY:
Inclusion Criteria:

1. Child is between 24 months to 36 months of age.
2. Singleton, full-term gestational birth (≥ 37 completed weeks of gestation), with a birth weight of ≥ 2.5 kg and ≤ 4.5 kg.
3. Healthy status based on medical history and physical examination
4. Weight- for-age and height-for-age within normal range on local childhood growth chart.
5. Written informed consent are obtained from both parents/legally authorized representative (LAR).
6. Parents/legally authorized representative must be able to provide evidence of the parental authority and identity.
7. Parents /legally authorized representative are of legal age of consent and must understand the informed consent and other study documents.
8. Parents/legally authorized representative are willing and able to fulfill the requirements of the study protocol.

Exclusion Criteria:

1. Known or suspected cows' milk protein intolerance / allergy, or lactose intolerance, or significant food allergies that impact a normal diet.
2. Prior to study participation, child has shown limited or no interest in drinking toddler milk.
3. Chronic infectious, gastrointestinal, metabolic, or genetic disease, including any disease/condition that impacts feeding or growth.
4. Use of systemic antibiotics or anti-mycotic medication in the 4 weeks preceding enrollment.
5. Child is currently consuming or has consumed any formulas or taking any supplement containing L. reuteri in the past 3 months.
6. Child is currently consuming or has consumed any formulas or taking any supplement containing GOS within the past 48 hrs prior to product in take, and who are not willing accept a temporary cessation of the consumption during the study period.
7. Child is currently participating in another investigational clinical trial.
8. Family or hierarchical relationships with the CIL team.

Ages: 24 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2023-04-06 (Actual); Study Completion 2023-04-06 (Actual)

PRIMARY OUTCOMES:
Colony forming units of feces (CFU/g) | Baseline (visit Day 0), Day 2, Day 3, Day4, Day 5, Day6 Day 7 and D21
  The primary end point is quantification of L. reuteri DSM 17938 in stool using quantitative polymerase chain reaction (qPCR).

SECONDARY OUTCOMES:
Gut microbiota | Between Day 0 and Day 21
  Diversity and functionality will be evaluated on at least 8 stools samples using shotgun metagenomic sequencing. Structure and prevalence of microbiota and evaluation of taxa and function in the survival of the probiotic.
Gastrointestinal (GI) tolerance and stooling patterns | Between Day 0 and Day 21
  Parent perceptions of GI symptoms and GI-related behaviors using Toddler Gut Comfort Questionnaire (GCQ) and stool frequency and consistency
Assessment of dietary variety | Between Day 0 and Day 21
  Dietary variety assessed using a parent-reported Food Frequency Questionnaire (FFQ)
Safety and tolerability | Between Day 0 and Day 21
  - Adverse events type, incidence, severity, and relationship to TEST1 and TEST2 products.

CONTACTS AND LOCATIONS:
Locations (1):
- Société des Produits Nestlé S.A., Lausanne, Canton of Vaud, Switzerland